CLINICAL TRIAL: NCT00243074
Title: A Phase II Trial of Novel Oral Anti-Angiogenic Agent AZD2171 (NSC-732208) in Malignant Pleural Mesothelioma
Brief Title: S0509 - AZD2171 in Treating Patients With Malignant Pleural Mesothelioma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02902; S0509; U10CA032102 (NIH); CDR0000446178 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2014-02

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is study how well AZD2171 works in treating patients with malignant pleural mesothelioma that cannot be removed by surgery. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective confirmed, complete, and partial response rates in patients with unresectable malignant pleural mesothelioma treated with AZD2171.

SECONDARY OBJECTIVES:

I. Determine the clinical benefit, in terms of objective response and stable disease rates, in patients treated with this drug.

II. Determine the 1-year median overall survival and progression-free survival in patients treated with this drug.

III. Determine the frequency and severity of toxic effects in patients treated with this drug.

IV. Correlate, preliminarily, pre- and post-treatment plasma vascular endothelial growth factor and soluble vascular cell adhesion molecule with clinical outcomes in patients treated with this drug.

V. Correlate, preliminarily, circulating endothelial cells with clinical outcomes in patients treated with this drug.

VI. Correlate variants of genes in the pathway targeted by this drug and variants of genes involved in the development of hypertension with the antiangiogenic property of this drug in these patients.

OUTLINE:

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial, sarcomatous, or biphasic malignant pleural mesothelioma

  * Unresectable disease

    * Residual disease after prior cytoreductive surgery allowed
* Measurable disease by CT scan or MRI
* Prior treatment with platinum-based chemotherapy required
* No known CNS metastasis
* Performance status

  * Zubrod 0-2
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* AST or ALT =< 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine =< 1.5 times ULN OR
* Creatinine clearance >= 50 mL/min
* Proteinuria =< 1+ by 2 consecutive dipstick tests taken >= 1 week apart
* No history of familial long QT syndrome
* Mean QTc =< 470 msec
* Systolic BP =< 150 mm Hg AND diastolic BP =< 100 mm Hg
* Must have New York Heart Association class I or II disease

  * Class II must be controlled with treatment
* Able to swallow and/or receive enteral medications via gastrostomy feeding tube
* Not requiring IV alimentation
* No active peptic ulcer
* No intractable nausea or vomiting
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in remission
* No history of hypersensitivity reaction to compounds of similar chemical or biological composition to the study drug
* Prior monoclonal antibody therapy targeting vascular endothelial growth factor (VEGF), VEGF receptor 1(VEGFR1) or VEGF receptor 2 (VEGFR2) allowed
* No other prior immunotherapy or biologic therapy
* No prior thymidine kinase inhibitor against VEGFR1 or VEGFR2
* No concurrent drugs or biologics with proarrhythmic potential
* No more than 1 prior chemotherapy regimen
* At least 28 days since prior chemotherapy (42 days for nitrosoureas or mitomycin) and recovered
* At least 21 days since prior radiotherapy and recovered
* At least 28 days since prior major surgery (e.g., thoracotomy or laparotomy) and recovered
* No prior surgery that would affect absorption
* Stable antihypertensive therapy allowed provided blood pressure (BP) parameters are met
* Concurrent enrollment on SWOG-S9925 allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Garland, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZD2171 (Cediranib Maleate)
Started | 54
Completed | 0
Not Completed | 54
Not completed — Ineligible | 6
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 36
Not completed — Death | 2
Not completed — not protocol specified | 1
Not completed — Did not receive any treatment | 1

BASELINE CHARACTERISTICS:
Population: Only eligible patients who received protocol treatment are included in the analysis. Of the 54 patients enrolled, 6 were ineligible and 1 addtional patients refused protocol treatment.
Arm/Group | AZD2171
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 66 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: confirmed complete and partial responses per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.".
Time Frame: Disease assessments for response were performed every 8 weeks for as long as the patient remained on protocol treatment, up to 5 years.
Population: Eligible patients who received any amount of AZD2171
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD2171 (Cediranib Maleate)
Number analyzed (Participants) | 47
percentage of participants | 9 [2 to 20]

2. Secondary Outcome: Overall Survival
Description: From the date of enrollment until the date of death due to any cause. Patients last known to be alive were censored at the date of last contact.
Time Frame: Daily during protocol treatment; then every 8 weeks until progression; then every 6 months for up to 3 years.
Population: Eligible patients who received AZD2171
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD2171
Number analyzed (Participants) | 47
months | 9.5 [5.6 to 10.7]

3. Secondary Outcome: Progression-free Survival
Description: From the date of enrollment until the date of disease progression (as determined by standard RECIST), symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free were censored at the date of last contact. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Every 8 weeks until disease progression or death, up to 5 years.
Population: Eligible patients who received AZD2171
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD2171
Number analyzed (Participants) | 47
months | 2.6 [1.7 to 3.7]

4. Secondary Outcome: Disease Control Rate
Description: The percentage of patients with a best of response of stable disease or better per standard RECIST. That is, patients whose best response was not increasing disease or death.
Time Frame: Every 8 weeks until disease progression progression, up to 5 years.
Population: Eligible patients who received AZD2171
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD2171
Number analyzed (Participants) | 47
percentage of participants | 44 [28 to 58]

5. Secondary Outcome: Objective Response Rate Per Modified RECIST for Pleural Tumors
Description: The sum of 6 pleural thickness measurements is added to sum of the longest diameters of all non-pleural measurable lesions. The resulting values are evaluated using RECIST.
Time Frame: Disease assessments for response were performed every 8 weeks as long as the patient remained on protocol treatment, up to 5 years.
Population: Eligible patients who received any amount of AZD2171
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD2171
Number analyzed (Participants) | 47
percentage of participants | 2 [0 to 11]

6. Secondary Outcome: Adverse Event Rates
Description: Adverse events per the NCI Common Toxicity Criteria version 3.0 that were possibly, probably or definitely related to protocol treatment. See adverse event tables for specific details.
Time Frame: Daily during protocol treatment
Population: All patients who received protocol treatment were assessed for adverse events. See adverse event tables for specific details.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2171 (Cediranib Maleate)
Number analyzed (Participants) | 47
Participants | 47

7. Secondary Outcome: Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Patients were assessed for adverse events every day for as long as they remained on protocol treatment, up to 5 years.
Population: Eligible patients who received any amount of protocol treatment with AZD2171 (cediranib maleate)
Measure: Number; unit: Participants
Arm/Group | AZD2171 (Cediranib Maleate)
Number analyzed (Participants) | 47
Participants
  Anorexia | 3
  Apnea | 1
  Ataxia (incoordination) | 1
  Cognitive disturbance | 1
  Colitis | 1
  Confusion | 2
  Constipation | 1
  Dehydration | 3
  Diarrhea | 4
  Dizziness | 1
  Encephalopathy | 1
  Fatigue (asthenia, lethargy, malaise) | 7
  Hypertension | 15
  Hypotension | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1
  Memory impairment | 1
  Metabolic/Laboratory-Other (Specify) | 1
  Muscle weakness, not d/t neuropathy - body/general | 1
  Nausea | 2
  Necrosis, GI - Esophagus | 1
  Neuropathy: sensory | 1
  Pain - Chest wall | 1
  Pain - Head/headache | 1
  Pain - Intestine | 1
  Pain - Pain NOS | 1
  Pain - Tumor pain | 1
  Perforation, GI - Ileum | 1
  Potassium, serum-low (hypokalemia) | 1
  Proteinuria | 2
  Rash: hand-foot skin reaction | 2
  Renal failure | 2
  Sodium, serum-low (hyponatremia) | 1
  Speech impairment (e.g., dysphasia or aphasia) | 1
  Thrombosis/thrombus/embolism | 3
  Vomiting | 1
  Weight loss | 2

ADVERSE EVENTS:
Time Frame: Daily during protocol treatment.
Arm/Group | AZD2171
Serious Adverse Events (participants affected / at risk) | 22/47
Other Adverse Events (participants affected / at risk) | 42/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2171 (N=47)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 1
Necrosis, GI - Esophagus (Gastrointestinal disorders) | 1
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1
Pain - Peritoneum (Gastrointestinal disorders) | 1
Perforation, GI - Colon (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Sudden death (General disorders) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 3
Infection-Other (Specify) (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Ataxia (incoordination) (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Hemorrhage, GU - Urethra (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2171 (N=47)
Hemoglobin (Blood and lymphatic system disorders) | 13
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 5
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 30
Distention/bloating, abdominal (Gastrointestinal disorders) | 5
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 17
Pain - Abdomen NOS (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 10
Constitutional Symptoms-Other (Specify) (General disorders) | 3
Edema: limb (General disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 35
Pain - Chest/thorax NOS (General disorders) | 6
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 8
AST, SGOT (Investigations) | 8
Alkaline phosphatase (Investigations) | 7
Creatinine (Investigations) | 9
Leukocytes (total WBC) (Investigations) | 3
Lymphopenia (Investigations) | 3
Metabolic/Laboratory-Other (Specify) (Investigations) | 9
Platelets (Investigations) | 7
Weight loss (Investigations) | 17
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 20
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 18
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 4
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 6
Pain - Neck (Musculoskeletal and connective tissue disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 5
Pain - Head/headache (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 3
Mood alteration - anxiety (Psychiatric disorders) | 4
Mood alteration - depression (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 14
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 5
Urinary frequency/urgency (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 18
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 17
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 34
Thrombosis/thrombus/embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less